CLINICAL TRIAL: NCT04005300
Title: Application of Prophylactic Low Calorie Feeding in Critically Ill Patients With High-risk Refeeding Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: refeeding syndrome
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness
Keywords: Refeeding syndrome; Enteral nutrition; Critical illness
MeSH Terms: conditions — Critical Illness; Refeeding Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low calorie feeding group (Experimental): Enteral nutrition was fed at 10-20kcal/kg/d for the first three days before identifying the refeeding syndrome
  Interventions: Dietary Supplement: restricted enteral nutrition
- standard calorie feeding group (Active Comparator): Enteral nutrition was fed at 500-750kcal/d for the first three days before identifying the refeeding syndrome
  Interventions: Dietary Supplement: standard enteral nutrition
- RFS group (No Intervention): The definition of RFS is that serum phosphate concentration decreased to below 0.87 mmol/L within 72 h after starting nutritional support and the biological variation needed to be greater than 30% decrease from any concentration previously recorded. And it is divided into three sub-group that is Group 1 that a drop of >0.16 mmol/L from any previous measurement, to below 0.65 mmol/L within 72 h after starting nutritional support, Group 2 that their serum phosphate concentration decreased to below 0.87 mmol/L within 72 h after starting nutritional support and the biological variation needed to be greater than 30% decrease from any concentration previously recorded, and Group 3 that their serum phosphate concentration decreased to below 0•32 mmol/L within 72 h after starting nutritional support.
- nRFS group (No Intervention): It is not up to the RFS definition

INTERVENTIONS:
Dietary Supplement: standard enteral nutrition — Enteral nutrition was treated within 48 hours after ICU and the calories were 500-750kcal/d
  Arms: standard calorie feeding group
Dietary Supplement: restricted enteral nutrition — Enteral nutrition was treated within 48 hours after ICU and the calories were 10-20kcal/kg/d for 3 days
  Arms: low calorie feeding group

SUMMARY:
Critically ill patients with high-risk nutrition are often at risk of refeeding syndrome(RFS), that the incidence of RFS is as high as 30-50%. It is sure that patients with refeeding syndrome were treated with restrictive enteral nutrition, but the definition of refeeding syndrome is not uniform, and there is still a lack of awareness high-risk patients of RFS to receiving early empirical low-calorie feeding intervention. So, we designed the study which is divided into three stages. Firstly, the monitoring rate of RFS was reviewed to evaluate the incidence of RFS in general ICU. Secondly, the best diagnostic criteria of RFS were prospectively defined. Finally, on this basis, it is assessed whether early low-calorie feeding could improve prognosis in high-risk patients with RFS.

DETAILED DESCRIPTION:
Stage 1: the monitoring rate of re-feeding syndrome in our department was reviewed to evaluate the incidence of re-feeding syndrome in severe patients,which is not described in detail; Stage 2:This part is a prospective observational study，divided into two group,that is, RFS group(their serum phosphate concentration decreased to below 0.87 mmol/L within 72 h after starting nutritional support and the biological variation needed to be greater than 30% decrease from any concentration previously recorded), which is divided into three sub-group(Group 1 that a drop of >0.16 mmol/L from any previous measurement, to below 0.65 mmol/L within 72 h after starting nutritional support, Group 2 that their serum phosphate concentration decreased to below 0.87 mmol/L within 72 h after starting nutritional support and the biological variation needed to be greater than 30% decrease from any concentration previously recorded, and Group 3 that their serum phosphate concentration decreased to below 0•32 mmol/L within 72 h after starting nutritional support.), and nRFS group(non-RFS that the serum phosphate do not up to the criteria). And the RFS group will be receiving the low-calorie feeding intervention, the nRFS group will be receiving the standard feeding according to the ASPEN guideline of 2016.

Stage 3: On this basis of stage 2, it is assessed whether early low-calorie feeding could improve prognosis in high-risk patients with RFS who was defined in NICE(National institute for the health and care excellence).The part of stage 3, divided into two groups that standard calorie feeding group and low calorie feeding group, aims to assess whether early low-calorie feeding could improve prognosis in high-risk patients with RFS.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients at least 18 years old;
* No history of enteral nutrition or parenteral nutrition within 1 week before ICU admission or ICU admission within 1 week;
* Mechanical ventilation patients requiring enteral nutrition support for >72h

Exclusion Criteria:

* refuse to join this study;
* enteral nutrition support for less than 3 days or have enteral nutrition contraindication;
* less than 18 years old;
* artificial nutrition (enteral/parenteral nutrition) has been applied to patients before admission;
* other factors of hypophosphatemia: continuous hemodialysis, recent parathyroidectomy, or hyperphosphatemia after treatment;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
The best diagnostic criteria for refeeding syndrome | 1 month mortality and the duration of mechanical ventilation
  Evaluate the best timing for intervention according to the lowest and the decline of serum phosphate
the incidence of refeeding syndrome | 3 day after treated with nutrition
  only according to serum phosphate standard

SECONDARY OUTCOMES:
duration of mechanical ventilation | 30 days
  The duration of mechanical ventilation in General ICU of our department in the same time admitted to ICU
survival rate | 28 days
  including discharge from hospital and ICU
occurrence of complications | 7 days
  including feeding intolerance, electrolyte disturbance

CONTACTS AND LOCATIONS:
Overall Officials: man huang, phD, Principal Investigator — Second affiliated hospital, Zhejiang university school of medicine; yunlong wu, master, Study Director — Second affiliated hospital, Zhejiang university school of medicine
Locations (1):
- Second affiliated hospital, Zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
One year after the article was published, and the opening lasted for one year
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the article was published, and the opening lasted for one year
Access Criteria: any study about refeeding syndrome
URL: https://pan.baidu.com/s/1nmmz9g9-cQrKkpJxVyglog

REFERENCES:
- [Background] Doig GS, Simpson F, Heighes PT, Bellomo R, Chesher D, Caterson ID, Reade MC, Harrigan PW; Refeeding Syndrome Trial Investigators Group. Restricted versus continued standard caloric intake during the management of refeeding syndrome in critically ill adults: a randomised, parallel-group, multicentre, single-blind controlled trial. Lancet Respir Med. 2015 Dec;3(12):943-52. doi: 10.1016/S2213-2600(15)00418-X. Epub 2015 Nov 18. PMID 26597128
- [Background] Rio A, Whelan K, Goff L, Reidlinger DP, Smeeton N. Occurrence of refeeding syndrome in adults started on artificial nutrition support: prospective cohort study. BMJ Open. 2013 Jan 11;3(1):e002173. doi: 10.1136/bmjopen-2012-002173. PMID 23315514
- See also: Restricted versus continued standard caloric intake during the management of refeeding syndrome in critically ill adults — http://linkinghub.elsevier.com/retrieve/pii/S2213-2600(15)00418-X
- See also: Occurrence of refeeding syndrome in adults started on artificial nutrition support — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3549252/